CLINICAL TRIAL: NCT04725955
Title: Postprandial Responses of Healthy Subjects to Wheat Bread Enriched With Encapsulated Hydroxytyrosol
Brief Title: Postprandial Responses to Hydroxytyrosol-enriched Bread
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Vaios T. Karathanos, Professor of Food Engineering and Physical Chemistry, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Harokopio_Hydroxytyrosol
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Postprandial Responses
Keywords: hydroxytyrosol; a-cyclodextrin; bread; glycaemic index; appetite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Glucose Solution (Placebo Comparator)
  Interventions: Other: Enriched wheat bread
- Wheat bread enriched with a-cyclodextrin (Active Comparator)
  Interventions: Other: Enriched wheat bread
- Wheat bread enriched with hydroxytyrosol encapsulated in a-cyclodextrin (Experimental)
  Interventions: Other: Enriched wheat bread
- White wheat bread (Placebo Comparator)
  Interventions: Other: Enriched wheat bread

INTERVENTIONS:
Other: Enriched wheat bread — Either 50g of glucose dissolved in 250mL water or white wheat bread or wheat bread enriched with 5mg a-cyclodextrin or wheat bread enriched with a 5mg mixture of a-cyclodextrin and encapsulated hydroxytyrosol (per 50g of available carbohydrates).

SUMMARY:
The amelioration of postprandial glucose and insulin responses to bread is of great importance since it may have significant beneficial effects on health. A number of studies have shown that hydroxytyrosol may have positive metabolic effects. However, this compound presents high hydrophilicity which constitutes the major barrier to its potential application in foods. Microencapsulation arises as a technological strategy to protect it and increase its stability. Alpha-cyclodextrin besides being a great carrier molecule, seems to also be beneficial to postprandial glucose levels. Enrichment of bread with encapsulated hydroxytyrosol could examine potential postprandial benefits.

Ten healthy normoglycemic subjects will participate in the study and will be provided with either a solution of glucose (reference food) or white wheat bread or wheat bread enriched with a-cyclodextrin or wheat bread enriched with hydroxytyrosol encapsulated in a-cyclodextrin, with 1-week intervals in amounts that yielded 50 g of available carbohydrates. Venous blood samples will be collected before consumption and at 30, 45, 60, 90, 120 and 180 min postprandially. Postprandial glucose, insulin and appetite-related hormone responses as well as glycemic index (GI) and subjective appetite ratings will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index
* Stable body weight for at least 3 months before enrollment
* Normal exercise, eating and drinking habits

Exclusion Criteria:

* Pregnancy and lactation
* Chronic medical illness (diabetes mellitus, cardiovascular disease, chronic liver, kidney, polycystic ovary syndrome or untreated thyroid disease)
* Use of nutritional supplements
* History of drug and/or alcohol abuse
* Psychiatric disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Glycaemic Index | Change between preprandial glucose measurements until 120 minutes postprandially
  Glycaemic Index of the enriched breads

SECONDARY OUTCOMES:
Insulin Response | Change between preprandial insulin measurements until 180 minutes postprandially
  Insulin Responses of the volunteers to the enriched breads (by a sandwich ELISA method, using a commercially available human insulin kit)
Appetite ratings | Change between preprandial subjective appetite measurements until 180 minutes postprandially
  Appetite ratings after the consumption of the enriched breads (evaluation of subjective appetite ratings, use of visual analogue scales)

CONTACTS AND LOCATIONS:
Locations (1):
- Laiko General Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Binou P, Stergiou A, Kosta O, Tentolouris N, Karathanos VT. Positive postprandial glycaemic and appetite-related effects of wheat breads enriched with either alpha-cyclodextrin or hydroxytyrosol/alpha-cyclodextrin inclusion complex. Eur J Nutr. 2022 Oct;61(7):3809-3819. doi: 10.1007/s00394-022-02913-z. Epub 2022 Jun 6. PMID 35668121